CLINICAL TRIAL: NCT05289388
Title: The Reliability of a Novel Index for Tissue Perfusion in Predicting Outcome in Patients With Septic Shock: a Prospective Observational Study.
Brief Title: a Novel Index for Tissue Perfusion in Predicting Outcome in Patients With Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Other Study IDs: N182022
Record Dates: First submitted 2022-03-13; First posted 2022-03-21 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lactate/CRT index — index will be calculated as the product of multiplying the CRT and serum lactate

SUMMARY:
Septic shock is a life-threatening condition with mortality rate of up to -40%. Septic shock is catheterized by altered microcirculation that leads to tissue hypoperfusion and ultimately multi-organ dysfunction. Hence, maintenance of adequate tissue perfusion is the mainstay of resuscitation of patients with septic shock.

Serum lactate is still considered the gold standard for evaluation of tissue perfusion. Thus, according to the latest definition, elevated serum lactate, as an indicator of tissue hypo-perfusion, is required for diagnosis of septic shock. However, lactate level change in response to resuscitation is slow even in survivors.

Capillary refill time (CRT) is a simple method for assessing peripheral perfusion. Monitoring CRT was found to be a good tool for guiding resuscitation and delayed CRT showed good ability in predicting mortality in patients with septic shock.

To the best of our knowledge, there is no previous report assessing the reliability of an index that include both serum lactate and CRT (lactate/CRT index) in predicting mortality in patients with septic shock.

We hypothesize that the lactate/CRT index would have good accuracy in predicting mortality in patient with septic shock.

DETAILED DESCRIPTION:
All patients will be monitored with; non-invasive and invasive arterial blood pressure, five-lead electrocardiography (ECG), hourly urinary output, and central venous pressure (CVP). Management of the patients will be done according to the latest surviving sepsis campaign guidelines in 2016. APACHE II score will be calculated on the time of admission using MDCalc ©.

Arterial blood gases, including serum lactate (blood gas analysis device GEM premier 300, Instrumentation Laboratory, Bedford, MA, USA), will be obtained at the time of intensive care unit admission, 6 and 12 hours after admission. Capillary refill time will be measured by applying enough pressure to cause skin blanching to the ventral surface of the distal phalanx of right index finger and the pressure will be then maintained for 10 seconds. The time for return of the normal skin color will be registered with a stopwatch. CRT will be recoded at the same time point as the blood sample.

The change in serum lactate (∆ Lactate), and CRT (∆ CRT) will be calculated as the difference between each two-consecutive measurement. Lactate/CRT index will be calculated as the product of multiplying the CRT and serum lactate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically suspected septic shock, older than 18 years old

Exclusion Criteria:

* Patients less than 18 years.
* patients with evident blood loss.
* patients with metastatic cancer.
* Patients with Child B or C liver cirrhosis
* patients with estimated glomerulo filtartion rate less than 30 ml/min/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients with clinically suspected septic shock according to the latest definition of septic shock (sepsis-3) "hypotension in a patient with sepsis requiring vasopressor therapy to maintain mean arterial pressure above 65 mmHg despite adequate fluid resuscitation in addition to elevated serum lactate level (above 2 mmol/L)"
Sampling Method: Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
the ability of Lactate/CRT index in predicting patient's outcome | 6 hour after admission
  multiplying the CRT and serum lactate

SECONDARY OUTCOMES:
ability of Lactate/CRT index in predicting patient's outcome | 12 hours after admission
  multiplying the CRT and serum lactate
ability of Lactate in predicting patient's outcome | 6 and 12 hours after admission
  mg/dl
ability of CRT in predicting patient's outcome | 6 and 12 hours after admission
  Capillary refill time will be measured by applying enough pressure to cause skin blanching to the ventral surface of the distal phalanx of right index finger and the pressure will be then maintained for 10 seconds. The time for return of the normal skin color will be registered with a stopwatch
change in serum lactate | WITHIN 1 HOUR, 6 and 12 hours after admission
  the difference between each two-consecutive measurement
change in CRT | WITHIN 1 HOUR, 6 and 12 hours after admission
  the difference between each two-consecutive measurement

CONTACTS AND LOCATIONS:
Overall Officials: ahmed hasanin, Principal Investigator — Cairo University Kasr Alainy Faculty of Medicine
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
the protocol and data supporting this study will be available from the PI upon reasonable request